CLINICAL TRIAL: NCT03652298
Title: Effects of a Neuroscience-based Technique on Post-traumatic Stress Disorder Symptoms, Inflammation, and Survival in Cancer Patients Announced of a Palliative Disease Progression and Their Partners
Brief Title: Effects of a Neuroscience-based Technique on Cancer Patients Announced of a Palliative Disease Progression and Partners
Acronym: NeuroPrevPTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment and of study staff
Sponsor: Centre Oscar Lambret (Other)
Collaborators: SCALab UMR CNRS 9193 Université de Lille (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NeuroPrevPTSD
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer; Bladder Cancer; Prostate Cancer; Kidney Cancer; Advanced Sarcoma
Keywords: PTSD; Memory Structuring Intervention (MSI); Cancer; Vagal breathing
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Stress Disorders, Post-Traumatic; Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: prospective randomized
Who Masked: Investigator
Masking Description: The research assistant blind to group assignments is responsible to conduct the three follows-ups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): In the experimental group, participants will perform vagal breathing (VB), followed by the MSI, followed again by VB. The VB component will guide participants how to perform deep slow vagal breathing by inhaling and counting 1-5, holding their breath and counting 1-2, and exhaling and counting 1-5, during 2-5 minutes. The MSI component will teach participants to chronologically organize the segments of their memory of the incurable diagnosis, to verbally label feelings or somatic sensations they had at that moment, and to provide causal links between the event's segments and causality to their feelings and sensations, following the protocol of Gidron et al. (2001).
  Interventions: Other: Memory structuring intervention + Vagal breathing
- Control Arm (Other): Participants in the control group will receive support and attention (usual care) and will be invited to recall announcement of the incurable disease progression. More precisely, they will be invited to express their associated thoughts and feelings, being free to talk about their experience, and the psychologist will react with empathy and support.
  Interventions: Other: support and attention (usual care)

INTERVENTIONS:
Other: Memory structuring intervention + Vagal breathing — The MSI component will teach participants to chronologically organize the segments of their memory of the incurable diagnosis, to verbally label feelings or somatic sensations they had at that moment, and to provide causal links between the event's segments and causality to their feelings and sensations, following the protocol of Gidron et al. (2001).
  In the MSI part, the patient will talk, and the therapist will note the different event parts and their real timing. Each time the patient says a feeling or sensation, the therapist will ask to verbally elaborate and provide the cause of these feelings and sensations. Then, the therapist will retell the story in a chronological manner, with verbal titles and causes for feelings and sensations. Finally, the patient will be asked to retell the story in this structured manner, after being explained how to do so.
  vagal breathing (i.e., deep, paced breathing) is a way to increase HRV, and thus parasympathetic activation
  Arms: Experimental arm
Other: support and attention (usual care) — support and attention (usual care)
  Arms: Control Arm

SUMMARY:
The diagnosis and treatment trajectory of cancer can constitute a traumatic event because these can be perceived as sudden, catastrophic and life threatening. One common mental disorder following traumatic events is post-traumatic stress disorder (PTSD), described as reexperiencing of the event (e.g., having intrusive thoughts), having avoidance of trauma memories, emotional numbing, and experiencing hyperarousal symptoms. To date, and to the best of the investigator's knowledge, few studies have focused on PTSD in advanced cancer, but the existing data show that these patients are at risk for experiencing PTSD symptoms.

Among the early interventions for preventing PTSD in people confronted by traumatic events is group debriefing, the retelling of the event, receiving empathy and compassion, and being encouraged to express feelings. However, four meta-analyses found debriefing to be ineffective. A neuroscience-based and evidence-based alternative may be the Memory Structuring Intervention (MSI) that tries to shift trauma processing from a limbic, emotional and somatic level to a frontal-cortical, cognitive and verbal level of processing. The MSI tries to achieve this shift by teaching people confronted with traumatic events to chronologically organize the segments of the event, to verbally label feelings or somatic sensations rather than re-experience them, and to provide causal links between the event's segments and causality to their feelings and sensations Since in males, sympathetic responses were more predictive of PTSD than in females , parasympathetic activation may be needed to be added to the MSI, for men. A main branch of the parasympathetic response is the vagus nerve, whose non-invasive index is Heart Rate Variability (HRV). One way to increase HRV, and thus parasympathetic activation, is through vagal breathing (i.e., deep, paced breathing). Therefore, adding to the MSI deep vagal breathing (VB) to reduce sympathetic hyperactivity, may increase connectivity between the amygdala and the frontal cortex. This may also increase the emotional regulation possibly yielded by the MSI, however in both genders.

The effects of the MSI + vagal breathing on PTSD symptoms and on prognosis in advanced cancer patients receiving announcement of terminal cancer have never been investigated. Furthermore, whether reduced inflammation and increased emotional regulation may account for such effects needs to be investigated at the fundamental level. This project reflects the merging of neuroscience, psychooncology and psychoneuroimmunology for better understanding and treating cancer patients, as well as their partners.

DETAILED DESCRIPTION:
Procedure for patients and partners:

Patients will be informed about the study by their treating oncologist at the end of the appointment, when they will be informed about the metastatic incurable progression of their disease (announcement visit). Oncologists will provide the patients a written description of the study, presenting the information previously orally provided by them, together with the consent form, to fill in. Signed informed consent will be sent back by post-mail if necessary (if participants ask for a time to think), using a pre-stamped envelope. Due to the objective to prevent distress, recruitment to the study and random assignment of the intervention need to be performed within the 7 days following this announcement visit, after making sure the patient is eligible for the study according to the inclusion and exclusion criteria.

Early after the announcement visit and consent collection, the clinical psychologist will call the patient before randomization in order to assess patients' level of stress from 1 (no stress) to 10 (maximal stress). Patients with a level higher or equal than 4 will be randomized in the study. For the patients with a stress level below or equal than 3, only background information will be collected in the study. These patients will receive the standard care.

Patients and their spouse will be randomly assigned together (i.e., if the spouse participates, he/she will be allocated to the same treatment arm as the patient) to receive the MSI + VB (experimental group) or to receive the supportive listening and attention (usual care serving as control condition), using an online centralized randomization program. Randomization will be implemented after the receipt of the consent form and balanced by (1) cancer type (bladder, prostate, kidney, colorectal cancer, sarcoma), (2) gender, as these two variables are identified as risk factors of PTSD (for cancer type) and as impacting the MSI effects (for gender) in the literature, and (3) the presence of the spouse during the announcement visit (yes/no), using a dynamic allocation program (minimization with a random factor set at 0.8).

For reasons of feasibility, no pre-screening aiming at including patients with a high risk of distress and potentially with high risk for developing PTSD will be realized. However, during the first telephone session, the psychologist will assess patients' level of stress using a 10-point likert scale, similar to a past study, before and after the MSI + VB intervention or the support and attention control session. This scale includes asking patients on a scale from 1 (no stress) to 10 (maximal stress) their level The treatment consists of a single telephone session conducted by a trained therapist maximum 10 days after receiving the announcement of the incurable disease progression. This is done in order to prevent PTSD, as was already done when the MSI treatment was developed in traffic accident survivors (Gidron et al., 2001, 2007). The same trained therapist will provide the MSI + VB intervention to the experimental group and give support and attention to the control group, in order to control for therapist's effects. This telephone session will be followed by 3 follow-up telephone assessments (a week, a month and 3 months after the previous telephone session), for collecting data by a research assistant who will not know in which group the participants are. All the sessions and interviews of the patient and his/her spouse (for treatments and for follow-up measures) will be conducted separately, and the information will remain confidential between the patient and the spouse. Each of these telephone calls will be conducted from the participating center, in order contact details of the participants remain inside the medical center to ensure the confidentiality of the data.

Experimental intervention. In the experimental group, participants will perform vagal breathing (VB), followed by the MSI, followed again by VB. The VB component will guide participants how to perform deep slow vagal breathing by inhaling and counting 1-5, holding their breath and counting 1-2, and exhaling and counting 1-5, during 2-5 minutes. The MSI component will teach participants to chronologically organize the segments of their memory of the incurable diagnosis, to verbally label feelings or somatic sensations they had at that moment, and to provide causal links between the event's segments and causality to their feelings and sensations, following the protocol of Gidron et al. (2001). In the MSI part, the patient will talk, and the therapist will note the different event parts and their real timing. Each time the patient says a feeling or sensation, the therapist will ask to verbally elaborate and provide the cause of these feelings and sensations. Then, the therapist will retell the story in a chronological manner, with verbal titles and causes for feelings and sensations. Finally, the patient will be asked to retell the story in this structured manner, after being explained how to do so.

patients in the MSI + VB group will be encouraged to perform it daily, for 5-10min, and especially before going to bed, to reduce any sleeping arousal associated with PTSD symptoms

Control. Participants in the control group will receive support and attention (usual care) and will be invited to recall announcement of the incurable disease progression. More precisely, they will be invited to express their associated thoughts and feelings, being free to talk about their experience, and the psychologist will react with empathy and support.

At Baseline for both arms, i.e., at the beginning of the telephone interview where the trained therapist will call the participants, the therapist will collect background information including age, gender, years of education, self-reported length of couple relationship and psychotropic medication (anxiolytic, antidepressant) in order to control the association between PTSD symptoms and anxiety and/or depressive disorder.

1. PTSD symptoms will be assessed by the post-traumatic checklist for DSM 5 (PCL-5; Weathers et al., 2013, French translation and validation by Ashbaugh et al., 2016).
2. Emotional regulation will be assessed by the BACQ scale (Finset et al., 2002).
3. Quality of life will be assessed by the EuroQol-5D scale (EQ-5D 3L)

In both groups, the trained therapist will also evaluate the degree of "natural" structuring regarding the way in which the patients/partners talk about the announcement visit. More precisely, the trained therapist will rate both groups on their level of chronological organization of their story from 1 = totally disorganized; 2 = a bit organized; 3 = chronologically very organized (in the MSI + VB group: before and after the MSI training; in the control group: at the first time they recall their story)

Afterwards, three follows-ups will be conducted by telephone: 1 week, 1 month and 3 months after the first intervention or control phone session.A research assistant blind to group assignments will collect the same self-reported measures initially collected by telephone at the first phone meeting. In sum, levels of PTSD symptoms and quality of life will be assessed at each time (initial phone meeting, 1 week, 1 month and 3 months). However, emotional regulation will be assessed at the first phone meeting and at one month only, in order to reduce patients' burden.

Patients and partners will also be asked if they have talked about the event, to recall how and how often they have spoken about the event since the last phone call.

For all the groups, medical information including type and stage of cancer and type of cancer treatments will be collected at baseline by the medical staff (as summarized in the table below). Levels of albumin and levels of C-reactive protein (CRP, reflecting inflammation) will also be obtained at baseline, 1 month and 3 months when patients will come in any case to the hospital for their medical appointments (no medical appointment is anticipated at 1 week, hence the absence of CRP and albumin measures at this time). Survival time will be monitored for all patients as well until the final analysis. We will calculate the quality-adjusted life years (QALY) for all patients, to reflect both quantity and quality of survival. This will be done using the length of survival weighted by patients' score on the EQ-5D scale.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged over 18 years old;
* Who received in the last 7 days the diagnosis of metastatic incurable bladder, prostate, kidney, colorectal or sarcoma cancer (including recurrence) during the announcement visit;
* Whose life expectancy is estimated ≥ 6 months by their treating oncologist;
* Who have a WHO performance score < 3 (to be coherent with the life expectancy);
* Who have an albumin level > 30g/liter (patients with an acceptable state of nutrition);
* Who gave their signed consent to participate in the study;
* Who are covered by a social insurance.

Exclusion Criteria:

* Patients diagnosed with cerebral metastases;
* Patients with locally advanced cancer without metastases;
* Patients with an advanced or metastatic cancer amenable to curative intent treatment;
* Patients suffering from a psychological vulnerability that might alter their reasoning or judgment capacities;
* Patients with a psychological or physical incapacity to answer the questionnaires, attested by the medical staff;
* Patients under custodial sentence or under tutelage or protection of vulnerable adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
PCL-5 score measurement at at 3 months (+/- 2 weeks) by the patient | 3 months
  PCL-5 means PTSD Checklist for DSM-5. This self-report rating scale assesses the presence and severity of PTSD symptoms. It includes 20 items. Each item is rated on a 0 (not at all) to 4 (extremely) response scale. The total score (0-80) is obtained by summing the scores for each of the 20 items. This total score reflects the severity of PTSD symptoms, and a cut-off of 32 reflects probable PTSD.

SECONDARY OUTCOMES:
Evolution of PCL-5 score in the first 3 months in the patient | 3 months
  Comparison of the PCL-5 score (PTSD symptoms severity score obtained by summing the scores for each of the 20 items) at 1 week, 1 month and 3 months after the first intervention.
  PCL-5 means PTSD Checklist for DSM-5. This self-report rating scale assesses the presence and severity of PTSD symptoms. It includes 20 items. Each item is rated on a 0 (not at all) to 4 (extremely) response scale. The total score (0-80) is obtained by summing the scores for each of the 20 items. This total score reflects the severity of PTSD symptoms, and a cut-off of 32 reflects probable PTSD.
The quality of life (QoL) score of the patient: EQ-5D | 3 months
  EQ-5D essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his health state in each of the dimensions. This decision results into a 1-digit number (number 1, 2, or 3) that expresses having no problems for 1, having some problems for 2, and having extreme problems for 3. The digits for the five dimensions is combined into a 5-digit number that describes the patient's health state, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Quality-adjusted life years (QALY) of the patient | 3 months
  QALY is the Quality-adjusted life years. This outcome will be calculating using the EQ-5D score and the survival time ,in order to take into account both the quantity and quality of life generated by an intervention. One QALY equates to one year in perfect health. If an individual's health is below this maximum, QALYs are accrued at a rate of less than 1 per year. To be dead is associated with 0 QALYs.
Inflammation level in the patients | 3 months
  Inflammation level will be assessed using CRP and albumin level
Emotion regulation in the patients | 3 months
  Emotion regulation evaluated by the BACQ scale. BACQ scale is the Brief Approach/Avoidance Coping Questionnaire.The scale contains 12 items based on a 5-point Likert scale ranging from 1 " Strongly disagree " to 5 "Totally agree ". The total score is calculated by the sum of the items (ranging from 12 to 60). It is also possible to calculate three subscores (i.e., approach index; resignation and withdrawal index; diversion index). The higher the total score, the more the participant use an approach coping.
Overall survival of the patients | 3 months
  Overall survival from randomization
PCL-5 score improvement in the partner | 3 months
  Improvement of the PCL-5 score at 3 months compared to Baseline. PCL-5 means PTSD Checklist for DSM-5. This self-report rating scale assesses the presence and severity of PTSD symptoms. It includes 20 items. Each item is rated on a 0 (not at all) to 4 (extremely) response scale. The total score (0-80) is obtained by summing the scores for each of the 20 items. This total score reflects the severity of PTSD symptoms, and a cut-off of 32 reflects probable PTSD.
PCL-5 score evolution in the partner | 3 months
  Evolution of PCL-5 score in the first 3 months, especially at 1 month. PCL-5 means PTSD Checklist for DSM-5. This self-report rating scale assesses the presence and severity of PTSD symptoms. It includes 20 items. Each item is rated on a 0 (not at all) to 4 (extremely) response scale. The total score (0-80) is obtained by summing the scores for each of the 20 items. This total score reflects the severity of PTSD symptoms, and a cut-off of 32 reflects probable PTSD.
Quality of life of the partner: EQ-5D scale | 3 months
  EQ-5D essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his health state in each of the dimensions. This decision results into a 1-digit number (number 1, 2, or 3) that expresses having no problems for 1, having some problems for 2, and having extreme problems for 3. The digits for the five dimensions is combined into a 5-digit number that describes the patient's health state, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Emotion regulation | 3 months
  Emotion regulation evaluated by the BACQ scale. BACQ scale is the Brief Approach/Avoidance Coping Questionnaire.The scale contains 12 items based on a 5-point Likert scale ranging from 1 " Strongly disagree " to 5 "Totally agree ". The total score is calculated by the sum of the items (ranging from 12 to 60). It is also possible to calculate three subscores (i.e., approach index; resignation and withdrawal index; diversion index). The higher the total score, the more the participant use an approach coping.

CONTACTS AND LOCATIONS:
Overall Officials: Georges-Michel REICH, MD, Principal Investigator — Centre oscar Lambret de Lille
Locations (1):
- Centre Oscar Lambret, Lille, France